CLINICAL TRIAL: NCT03701113
Title: Evaluation of a Milk-Based Protein Supplement to Effect a Positive Change in Bone Health in Post-Menopausal Women Aged 50 to 70 y at Risk of Osteoporosis
Brief Title: Milk Protein and Bone Health in Postmenopausal Women
Acronym: OSTEOMILK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: Dairygold Cooperative Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018_04_05_EHS
Record Dates: First submitted 2018-09-28; First posted 2018-10-09 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Bone and Bones; Osteoporosis Risk; Osteoporosis, Postmenopausal
Keywords: Osteoporosis; Postmenopausal; Bone Turnover Markers; Dairy Products
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Intervention Model Description: A block randomised, controlled study among healthy, post-menopausal women with osteopenia receiving a milk-based protein supplement (MBPS) in the evening, or not (CONTROL), for a period of 24 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Milk-based protein matrix (MBPM) (Active Comparator): Intervention: Dietary Supplement : Test Product Intervention: Diagnostic Test : Aerial Bone Mineral Density (BMD) Intervention: Diagnostic Test : Bone Turnover Composition of Test Product - 25g of milk-based proteins + 1000mg dairy-based calcium fortified with 40ug Vit D flavoured and textured supplied food grade and product tested by Dairygold Co-operative Society, Mitchelstown, Ireland.
  Interventions: Dietary Supplement: Milk-based protein matrix (MBPM)
- CONTROL (Other): Intervention: Habitual dietary behaviour Intervention: Diagnostic Test : Aerial Bone Mineral Density (BMD) Intervention: Diagnostic Test : Bone Turnover
  Interventions: Dietary Supplement: Habitual dietary behaviour

INTERVENTIONS:
Dietary Supplement: Milk-based protein matrix (MBPM) — Ingestion of the Test Product at 10:00 pm, post-absorptive of the evening meal, each day for the 24 week period of intervention
  Arms: Milk-based protein matrix (MBPM)
Dietary Supplement: Habitual dietary behaviour — Subjects to maintain habitual dietary behaviour for the 24 week intervention
  Arms: CONTROL

SUMMARY:
The process of bone remodeling exhibits pronounced diurnal pattern that is important for bone health. A balanced rate of bone resorption is required to maintain bone health, a balance that can be disturbed during the life-cycle to effect net rate of formation (as occurs during growth and development to adulthood) or net resorption (as occurs, for example, during the menopause). Bone turnover is a nutritionally modulated process and the investigators believe a milk-based protein supplement (MBPS) can modulate beneficially the rate of bone resorption over the time period when bone remodeling is most active i.e. late evening/overnight. In this novel approach to the timing of nutrient ingestion, the proposed nutrient intervention seeks to modify (reduce) the rate of bone resorption and promote the rate of bone formation to the benefit of bone health in this at risk population..

DETAILED DESCRIPTION:
Study design:

A block randomised, controlled study among healthy, post-menopausal women with osteopenia receiving a milk-based protein supplement (MBPS) in the evening, or not,(CONTROL) for a period of 24 weeks.

Composition of MBPM - 25g of milk-based proteins + 1000mg dairy-based calcium fortified with 40ug Vit D flavoured and textured. All formulations to be supplied food grade and product tested by Dairygold Co-operative Society, Mitchelstown, Ireland.

Participants:

60 Post-menopausal women with osteopenia as determined by site-specific bone mineral density BMD (DXA) diagnosed and screened by a clinician and for dietary intake of calcium and Vit D by a clinical dietitian.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women aged 50-70y. Assessed by site-specific BMD to be osteopenic. Assessed by clinical screen to be otherwise healthy and free from other illness or current medication likely to influence the study outcome.

Exclusion Criteria:

* Intolerance to dairy-based food products

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Aerial Bone Mineral Density (BMD) | Change from Baseline BMD at 24 weeks
  Site specific (hip and lumbar) BMD measured by Dual Energy X-ray Absorptiometry (DXA)

SECONDARY OUTCOMES:
Bone Resorption | Change from Baseline CTX, NTX and DPD at 24 weeks
  Measured by biomarkers of bone resorption in fasting blood, i.e. C-terminal telopeptide of type I collagen (CTX, ng/ml), and diurnal (24h) urinary deoxypyridinoline (DPD, nmol/mmol creatinine) and N-terminal telopeptide of type I collagen (NTX, nmol/mmol creatinine) excretion normalised for urinary creatinine.
Bone Formation | Change from Baseline P1NP at 24 weeks
  Measured by a biomarker of bone formation in fasting blood, i.e. serum pro-collagen type 1 N-terminal propeptide (P1NP, ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Jakeman, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Center for Interventions in Inflammation Infection and Immunity — http://ul.ie./4i
- Available data/document: Study Protocol: 2018_04_05_EHS — http://www.ul.ie/ehs/research-ethics — Contact The EHS Research Ethics Contact Point of the Education and Health Sciences Research Ethics Committee, Room E1003, University of Limerick, Limerick, Ireland

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT03701113/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT03701113/SAP_001.pdf